CLINICAL TRIAL: NCT00264706
Title: PolyArginine Treated vEiN grafTs (PATENT)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Reformulation of test compound
Sponsor: Lumen Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Lumen-01-CS-1
Record Dates: First submitted 2005-12-11; First posted 2005-12-13 (Estimated); Last update posted 2016-09-08 (Estimated); Status verified 2016-09

CONDITIONS: Saphenous Vein Graft Disease
MeSH Terms: interventions — nonaarginine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (1):
- Participant (Other): Internal control study
  Interventions: Drug: Nona-L-arginine

INTERVENTIONS:
Drug: Nona-L-arginine

SUMMARY:
The primary objectives of this trial are: 1) to evaluate the safety of NONA-L-ARGININE in ex vivo application to saphenous vein segments prior to grafting; and, 2) to obtain preliminary data on the biological effects of NONA-L-ARGININE, as compared to placebo, in the prevention of neointimal hyperplasia.

DETAILED DESCRIPTION:
LT-1951 is an aqueous solution of NONA-L-ARGININE. The drug efficiently penetrates into vascular tissues like the saphenous vein and supplies the tissue with a sustained reservoir of L-arginine, the substrate for production of nitric oxide. Nitric oxide (NO) is an important vasoactive and cell signaling compound implicated in suppression of neointimal hyperplasia. NO limits neointimal hyperplasia by inhibiting monocyte chemotaxis and adherence, platelet adherence and aggregation, and vascular smooth muscle cell proliferation.

A dramatic reduction of neointimal hyperplasia following treatment with LT-1951 has been demonstrated in preclinical vein to artery interposition studies in several animal models. Marked improvement following a single ex vivo application of LT-1951 in interposition grafts demonstrated that the beneficial effect of the drug is not dependent upon continued treatment of the grafted tissue.

In the PATENT trial, saphenous vein grafts are harvested in the usual manner from the patient's leg and are bathed in LT-1951 or placebo ex vivo (at normal pressure and temperature) before being rinsed and implanted into the patient. Because LT-1951 is applied only to the graft, there is minimal systemic exposure and risk to the patient.

All patients in this study will receive treatment with both NONA-L-ARGININE and vehicle control. This within-patient, placebo-controlled, study will be double-blinded and randomized. For each patient, one of the comparable vein grafts will receive treatment with placebo, while the other will receive treatment with NONA-L-ARGININE. Any third vein graft used in the procedure will be treated as per the first vein graft, while any fourth vein graft will be treated as per the second vein graft.

The first cohort of 20 patients will be the primary safety subgroup. This subgroup will be evaluated in combination with a second cohort of 30-80 patients for assessment of efficacy endpoints. During follow-up, all patients will have clinical visits at 6 weeks, which will include Computed Tomographic Angiography (CTA). Patients will undergo Intravascular Ultrasound-coronary angiography (IVUS-angio) at 12 months and optional CTA at 6, 12 and 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be 35-85 years of age and able to give informed consent.
2. Coronary artery disease requiring bypass grafting using at least two saphenous vein bypass grafts carried out through median sternotomy and utilizing cardiopulmonary bypass.
3. Use of an approved statin anticipated for at least 24 months after surgery.
4. Subject must not be a candidate for concurrent ventricular surgical restoration, AICD placement, or valvular surgery.
5. Agreeable to CTA at 6 weeks and IVUS intervention at 12-months post-CABG. Subjects agreeable to additional CTA at 6, 12 and 24 months preferred.

Exclusion Criteria:

1. Acute traumatic injury or vasculitis.
2. Insulin-dependent diabetes.
3. Procedure is for revision for an existing bypass graft.
4. Procedure is to be minimally invasive (except for harvesting of the graft segment).
5. Concurrent cardiac valvular surgery.
6. Patients with any medical condition that, in the investigator's judgment, makes the patient ineligible or places the patient at undue risk (e.g. conditions that preclude standard invasive follow-up procedures such as IVUS and angiography, i.e. renal failure, bleeding diathesis, or peripheral vascular disease preventing catheterization via the groin).
7. Subject has clinical evidence of infection that the Investigator deems significant to the completion of the procedure, or that could compromise the subject's safety.
8. Subject has recent history (within past 6 months) of alcohol or drug abuse.
9. If female, subject is pregnant or trying to become pregnant.
10. Calculated creatinine clearance < 30 mls/min for non-diabetics or < 50 mls/min for non-insulin dependent diabetics.

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2005-03; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Safety - as assessed by the nature and frequency of clinical adverse event at 6 weeks post-surgery. | 6 weeks
Efficacy - Volume obstruction of the vein grafts measured by IVUS at 1 year. | 1 year

SECONDARY OUTCOMES:
1. Volume obstruction adjacent to the proximal and distal anastomoses, and within the body of the graft; 2. Intima:media ratio; 3. Minimal and maximal luminal diameter; and, 4. lumen volume:vessel volume. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Brister, M.D., Principal Investigator — Toronto General Hospital
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada

REFERENCES:
- See also: Click here for additional information on Saphenous Vein Graft Disease and the PATENT study. — http://www.lumentherapeutics.com/page/clinical.htm